CLINICAL TRIAL: NCT06853366
Title: Validation of the Short Form of the "Lower Urinary Tract Symptoms Treatment Constraints Assessment" Questionnaire
Acronym: FC-LUTS-TCA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0031_LUTS-TCA
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Urologic Disorders
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
For many years, the evaluation of treatments has been a central issue in patient care. The various domains assessed have gradually evolved over time, ranging from satisfaction, improvement and quality of life, to the more recent introduction of the Patient Reported Outcome Measure (PROM). These questionnaires or measurement scales (PROMs) focus assessment on the patient and his or her direct experience. Statistical validation of numerous assessment tools has made it possible to quantify objectively many areas of assessment that were initially linked to the patient's feelings, and therefore to their subjectivity. Thus, improvement, quality of life, patient expectations and goal attainment have been the preferred areas for the development of these PROMs.

However, certain areas have been sidelined in the creation of these tools. For example, the constraint of care or the side effects or negative effects of care have not been studied through specific means of evaluation.

In response to this shortcoming, we have developed a questionnaire specifically designed for neuro-urological treatments in a neurological patient population.

The LUTS-TCA (Lower Urinary Tract Symptoms Treatment Constraints Assessment) was developed in French and statistically validated in 2019.

The aim of the study is to create a short form of the LUTS TCA in French, in a population of neurological patients.

This short form, which would be easier to use and interpret, would simplify its use in everyday practice. Indeed, a large majority of neuro-urology patients suffer from neurodegenerative or progressive pathologies, marked by significant and disabling physical and psychological fatigue symptoms. Long-form questionnaires, or the addition of multiple assessment questionnaires during a single visit to the department, make overall assessment more complex.

In addition, this short-form questionnaire is presented in a slightly different form to the long-form version, showing several domains of constraint (physical, social, psychological and care system). This classification should simplify the interpretation and understanding of care constraint, by and for patients.

For the patient, the validation study will take place in 2 phases:

* A first phase at the time of the consultation (Day 0): response to the questionnaires making up the study, i.e. the short form of the LUTS TCA (appendix 2), then the validated form of the LUTS TCA (22 questions) and finally the PGI (two questions).
* A second phase, at a distance from the consultation (Day 14 post-consultation): response to the short form of the LUTS TCA (questionnaire handed out at the consultation, accompanied by a stamped envelope for return).

DETAILED DESCRIPTION:
For many years, the evaluation of treatments has been a central issue in patient care. The various domains assessed have gradually evolved over time, ranging from satisfaction, improvement and quality of life, to the m ore recent introduction of the Patient Reported Outcome Measure (PROM). These questionnaires or measurement scales (PROMs) focus assessment on the patient and his or her direct experience. Statistical validation of numerous assessment tools has made it possible to quantify objectively many areas of assessment that were initially linked to the patient's feelings, and therefore to their subjectivity. Thus, improvement, quality of life, patient expectations and goal attainment have been the preferred areas for the development of these PROMs.

However, certain areas have been sidelined in the creation of these tools. For example, the constraint of care or the side-effects or negative effects of treatment have been little studied using specific assessment tools.

In the field of neurology or neuro-urology, only a few multidimensional questionnaires take these domains into account. The main one is Qualiveen, which, in addition to quality of life, looks at discomfort, constraint, fear and patient experience. Other questionnaires, less specific in terms of population, enable a multidimensional evaluation of treatments according to 4 domains (efficacy, side effects, ease of use and overall satisfaction) for the Treatment Satisfaction Questionnaire for Medication (TSQM) or 6 domains (side effects, efficacy, practical aspects of drug treatment, effects of drug treatment on daily life, medical follow-up and overall opinion of treatment) for the Treatment Satisfaction with Medicine Questionnaire (SatMed-Q). These 2 multi-dimensional questionnaires do not allow for a targeted assessment of the constraint of care, which represents a much broader domain than the simple side effect or ease of use of a treatment. What's more, a mixed assessment, both positive (improvement, efficacy) and negative (side-effects) on the same questionnaire, may well limit the interpretation of results and patient understanding.

In response to this shortcoming, a specific treatment constraint questionnaire has been developed for neuro-urological treatments in a neurological patient population.

The LUTS-TCA (Lower Urinary Tract Symptoms Treatment Constraints Assessment) was developed in French and statistically validated in 2019. This 22-item questionnaire provides a general assessment of therapeutic constraint (physical, social, psychological, etc.). The "detailed" study of therapeutic stress is an important part of the overall therapeutic assessment of these neurological patients, as therapeutic management is often multiple and complex in terms of treatments, examinations, follow-up and impact on daily life.

The use of specific, validated tools to take account of care constraints is important, and is just as justified as the assessment of satisfaction or therapeutic improvement.

The "detailed" study of care constraints is an important part of the overall therapeutic assessment of these neurological patients, as therapeutic management is often multiple and complex in terms of treatments, examinations, follow-up and impact on daily life.

The use of specific, validated tools to take account of care constraints is important, and is just as justified as the assessment of satisfaction or therapeutic improvement.

One of the most widely used questionnaires for measuring treatment improvement is the Patient Global Impression of Improvment (PGI-I). The PGI-I takes the form of a single question, with a 7-level Likert scale ranging from +3 (much improved) to -3 (not improved at all). These positive and, above all, negative levels can be confused with the care constraint for the negative part of the response mode. To avoid measuring the same thing twice (negative PGI-I and LUTS TCA), it is vital to be able to measure the 2 parameters independently.

The aim of the study is to create a short form of the LUTS TCA in French, in a population of neurological patients.

This short form, which would be easier to use and interpret, would simplify its use in everyday practice. Indeed, a large majority of neuro-urology patients suffer from neurodegenerative or progressive pathologies, marked by significant and disabling physical and psychological fatigue symptoms. Long-form questionnaires, or the addition of multiple assessment questionnaires during a single visit to the department, make overall assessment more complex.

In addition, this short-form questionnaire is presented in a slightly different form to the long-form version, showing several domains of constraint (physical, social, psychological and care system). This classification should simplify the interpretation and understanding of care constraint, by and for patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Patients with central or peripheral neurological pathology, followed and managed for vesico-sphincter disorders
* Patients receiving urinary treatment for more than 3 months
* No therapeutic modification between D0 and D14 of the questionnaire
* French-speaking patients (able to read, write and understand French)

Exclusion Criteria:

* Minor patients (age ≤ 17 years)
* Patients who have stopped urinary treatment
* Patients with major cognitive impairment
* Patients who speak little or no French
* Patients who refused to participate in research, or who objected to the use of their data for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in the urology department of the Casanova and Pitié Salepêtrière Hospital
Sampling Method: Non-Probability Sample
Enrollment: 242 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Demographic data | day 1
  Age
Demographic data | day 1
  sex
Mecical history | day 1
  The medical history of the patient (treatement, diseases, diagnosis...)
Treatment(s) | day 1
  Treatment(s) taken by the patient (starting date, dosage, end date (if available)...)
LUTS- TCA Questionnaire (short form) | day 1
  This questionnaire only has one question.
LUTS-TCA questionnaire (original) | day 1
  The answers provided by this questionnaire (22 items)
PGI questionnaire | day 1
  The answers of the PGI questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - La pitié salpêtrière, Paris, paris
  - Casanova Hospital, Saint-Denis, Seine saint denis